CLINICAL TRIAL: NCT04392843
Title: Effect of Fasting on Insulin-induced Hypoglycemia Counterregulation in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jason Winnick, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-0625
Record Dates: First submitted 2020-05-08; First posted 2020-05-19 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Hypoglycemia
Keywords: glucagon; hepatic glucose production; liver glycogen
MeSH Terms: conditions — Hypoglycemia | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Two subjects will undergo two metabolic studies, one after having remained fasted and one after having eaten breakfast and lunch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (Other): Subjects will remain fasted prior to insulin-induced hypoglycemia.
  Interventions: Other: Fasting
- Feeding (Active Comparator): Subjects will eat a normal breakfast and lunch prior to insulin-induced hypoglycemia.
  Interventions: Other: Feeding

INTERVENTIONS:
Other: Fasting — Subjects remain fasted prior to insulin-induced hypoglycemia.
  Arms: Fasting
Other: Feeding — Subjects eat a normal breakfast and lunch prior to insulin-induced hypoglycemia.
  Arms: Feeding

SUMMARY:
Iatrogenic hypoglycemia is still considered to be the number one barrier to effective glycemic control in patients with type 1 diabetes (T1D). In a previous study, we observed in dogs that liver glycogen content can be a determinant of hormonal and hepatic responses to insulin-induced hypoglycemia. In the experiments described herein, we will determine if nutritionally-manipulated changes in liver glycogen concentrations have an impact on hypoglycemic counterregulation in non-T1D control subjects.

DETAILED DESCRIPTION:
Because patients with type 1 diabetes (T1D) are required to estimate and administer their own insulin requirements, they frequently overestimate their needs. This often leads to debilitating insulin-induced hypoglycemia, which is the number one barrier to the safe, effective management of glycemia in this population. In addition to the difficulty estimating one's own insulin requirements after a meal, counterregulatory hormone responses to hypoglycemia are impaired in patients with T1D, thereby reducing hepatic glucose production (HGP) and increasing the depth and duration of the hypoglycemic episode.

The discovery of ways by which counterregulatory responses to hypoglycemia can be improved is a priority. In previous experiments in the dog, we observed that experimentally decreasing liver glycogen content (using a 4-hour infusion of glucagon into the hepatic portal vein) reduces counterregulatory hormone secretion during insulin-induced hypoglycemia, thereby reducing hepatic glucose production (HGP). Interestingly, people with T1D have low fasting hepatic glycogen concentrations and the accretion of the sugar in the liver throughout the day is also diminished. Therefore, it is of great interest to understand the relationship between fasting, which would lower liver glycogen levels compared to normal caloric intake, and the counterregulatory responses to insulin-induced hypoglycemia. Furthermore, the translational significance of the investigator's previous findings is also of great importance. To these ends, the studies proposed herein will determine the effect of fasting on hypoglycemic counterregulation in healthy, non-T1D subjects. We hypothesize that fasting will diminish the hormonal and hepatic responses to insulin-induced hypoglycemia.

Each subject will undergo two trials; one where they eat an isocaloric breakfast and lunch prior to an insulin-induced hypoglycemic challenge and a second one during which they remain fasted prior to the hypoglycemic challenge. This study design will allow us to assess the relationship between fasting and the counterregulatory responses to insulin-induced hypoglycemia. For these preliminary studies, only healthy subjects will be studied, thereby reducing their complexity (e.g., no overnight inpatient visits or the need to adjust insulin doses during the feeding periods). Upon completion, we intend to study the more metabolically vulnerable T1D patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any race or ethnicity.
* Aged 21-40 years.
* Fasting glucose lower than 110 mg/dL.
* Non-obese (BMI <28 kg/m2).
* Otherwise healthy as determined by a physician (i.e., no acute or chronic conditions/ illnesses that might have an impact on the results of the study).

Exclusion Criteria:

* Pregnant women.
* Cigarette smoking.
* Taking inflammation-targeting steroids (e.g., prednisone).
* Taking medications targeting adrenergic signaling (e.g., beta-blockers, bronchodilators).
* Hematocrit less than 33%.
* Presence of HIV or hepatitis (due to their deleterious effects on the liver).
* The presence of cardiovascular or peripheral vascular disease.
* The presence of neuropathy, retinopathy or nephropathy.
* A diagnosis of diabetes (type 1 or type 2) or a detection of the presence of any other disease or condition by one of the study doctors, that would be expected to confound the responses to insulin-induced hypoglycemia or make participation in the study dangerous to the individual.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Glucagon | During intervention
  From plasma
Epinephrine | During intervention
  From plasma
Glucose infusion rate | During intervention
  Required to clamp glucose at 50 mg/dL

SECONDARY OUTCOMES:
Hepatic glucose production | During intervention
  From plasma
Peripheral glucose uptake | During intervention
  From plasma

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warner SO, Dai Y, Sheanon N, Yao MV, Cason RL, Arbabi S, Patel SB, Lindquist D, Winnick JJ. Short-term fasting lowers glucagon levels under euglycemic and hypoglycemic conditions in healthy humans. JCI Insight. 2023 Jun 22;8(12):e169789. doi: 10.1172/jci.insight.169789. PMID 37166980